CLINICAL TRIAL: NCT02058862
Title: Effects of a Superimposed Electrical Stimulation Knee Garment on Strength, Function, Inhibition, Cortical Excitability, and Patient Reported Outcomes After Knee Surgery
Brief Title: Effect of a Home-based Electrical Stimulation on Quadriceps Function After Knee Surgery
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Collaborators: DonJoy Orthopedics (Unknown)
Responsible Party: Principal Investigator, Caitin Conley, PhD, ATC, University of Kentucky
Other Study IDs: 13-0776-F2L
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Post-operative Quadriceps Weakness; Post-operative Quadriceps Inhibition; Adherence to Post-operative Treatment; Post-operative Lower Extremity Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if a home-based electrical stimulation (ES) program is more effective than the standard of care (SOC) at improving quadriceps function, functional outcomes, patient reported outcomes, and treatment compliance in patients recovering from knee surgery. It is hypothesized that there will be significantly better outcomes and compliance in ES group when compared to the SOC group.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of home-based neuromuscular electrical stimulation applied via a knee sleeve on strength, function, inhibition, and patient reported outcomes. Strength will be evaluated via isometric knee extension, neuromuscular inhibition will be assessed via a superimposed burst technique, and cortical excitability will be assessed via transcranial magnetic stimulation. In addition, we will evaluate function through a single-leg hop task, star excursion balance test, and a step down task. Patient reported outcomes will be assessed via the: Veterans Rand 12 Item Health Survey (VR-12), Knee Osteoarthritis Outcomes Score (KOOS), the International Cartilage Repair Society (ICRS), the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, and the Lysholm scale.

Once a participant is identified as eligible and consents to enroll in the study, they will be allocated to either an intervention or control group. The participants in the intervention group will receive a knee sleeve that has a neuromuscular ES unit embedded into the garment (EMPI Phoenix, DJO Global, Vista, California) in addition to SOC. A superimposed electrical signal (maximal toleration) will be utilized during treatment in order to successfully overload the muscle. During the electrical stimulation the participants will be instructed to perform an isometric contraction and hold this contraction through the length of the stimulation. Beginning one week post-operatively the participants will be instructed to perform NMES treatment 3 times a day for 20 minutes 5 times a week for 12 weeks. The stimulation will be delivered at a frequency of 75Hz with a duty cycle of 4 seconds on and 10 seconds off. The control group will be treated with the current SOC, performing a home-based treatment of volitional isometrics contractions without the addition of neuromuscular electrical stimulation beginning on the third day post-operatively. Participants will perform 20 isometric contractions holding each contraction for 10 seconds 3 times a day 5 times a week for 12 weeks. Participants will be instructed to keep a treatment log documenting at each session how many exercises and at what intensity they performed.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for surgery to address pain, injury, or dysfunction of the knee joint.
* Must be able to communicate using the English language

Exclusion Criteria:

* Previous surgery to the contralateral ankle, hip, or knee
* Injury to the hip, ankle, or contralateral knee in the past six months
* Currently being treated for low back pain
* Presence of a heart condition/pacemaker
* History and/or family history of seizures/epilepsy
* Vestibular or other balance disorders

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from the University of Kentucky Orthopaedics and Sports Medicine Clinic who are seeking surgical treatment for a disease/injury of the knee.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Isometric knee extension torque | Preoperative baseline, 1 month post-operative, 3-4 month post-operative, 6 month post-operative, and 12 month post-operative
  Knee extension torque derived from a maximal voluntary isometric contraction
Quadriceps activation | Preoperative, 3-4 month post-operative, 6 month post-operative, and 12 month post-operative
  Central activation ratio of the quadriceps derived from the superimposed burst technique

SECONDARY OUTCOMES:
Patient-reported outcomes | Preoperative, 1 month post-operative, 3-4 month post-operative, 6 month post-operative, and 12 month post-operative
  Patient-reported outcome measures will include the following: Veterans Rand 12 Item Health Survey (VR-12), Knee Osteoarthritis Outcomes Score (KOOS), the International Cartilage Repair Society (ICRS), the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, and the Lysholm scale
Functional outcomes | Preoperative, 3-4 month post-operative, 6 month post-operative, and 12 month post-operative
  Functional outcome measures will include the following: Single-leg hop, 30-second step down, and star-excursion balance test.
Cortical excitability | Preoperative, 1 month post-operative, 3-4 month post-operative, 6 month post-operative, and 12 month post-operative
  Individuals who have been diagnosed with epilepsy or have a family history of epilepsy may be at risk of seizure during cortical excitability testing. Therefore, these individuals will be excluded from this study. Otherwise, this measure is considered to be safe and is used in the realms of both medicine and research.

OTHER OUTCOMES:
Treatment compliance | Preoperative, 1 month post-operative, 3-4 month post-operative, 6 month post-operative, and 12 month post-operative
  The number and duration of treatments performed by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Conrad M Gabler, PhD, ATC, Principal Investigator — University of Kentucky; Caitlin E Whale Conley, PhD, ATC, Principal Investigator — University of Kentucky; Carl G Mattacola, PhD, ATC, Study Chair — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky Musculoskeletal Laboratory, Lexington, Kentucky
  - University of Kentucky Orthopaedics and Sports Medicine Clinic, Lexington, Kentucky